CLINICAL TRIAL: NCT01695512
Title: Open, Prospective, Multicenter Trial to Evaluate the Clinical Significance of Combined Serological (Galactomannan ELISA, 1->3-β-D Glucan Assay) and Molecular (Nested Aspergillus PCR Assay, Multifungal DNA Microarray) Diagnostic Assays to Detect and Characterize Fungal Pathogens in Bronchoalveolar Lavage (BAL) and Blood Samples of Hematological High Risk Patients and to Detect Point Mutations Conferring Azole Resistance
Brief Title: Diagnostic Study of Combined Biomnarker Testing in Bronchoalveolar Lavage Samples of Immunocompromised Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Heidelberg University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Dieter Buchheidt, Professor Dr. Dieter Buchheidt, Heidelberg University
Other Study IDs: University of Heidelberg; Grant Funding number (Other Grant/Funding Number: Gilead Sciences #PO 201 001 756)
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Invasive Aspergillosis; Acute Leukemia; Biomarkers; Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Only fungal DNA is retained and investigated
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Immunocompromised Patients: Patients with acute leukemia undergoing induction chemotherapy or undergoing allogeneic stem cell transplantation
- Control Group: Patients underdoing bronchoscopy and diagnostic BAL without immunosuppression and without signs of infection (Sarcoidosis, Lung Cancer)

SUMMARY:
The aim of our prospective and multicentre diagnostic study is therefore to elucidate on the sensitivity and specificity rates of these serologic markers in combination with molecular tools (both an Aspergillus specific and a multifungal PCR based assay), as serologic mark-ers are not pathogen-specific, and furthermore to define species-specific cut-off values for BDG in BAL samples.

Additionally, if genomic material of Aspergillus fumigatus is detected by PCR in a clinical sample, we investigate fungal DNA for point mutations in the cyp51A gene mediating resis-tance against common mould-active triazoles with novel rapid, sensitive and specific, non-culture-based PCR-assays and sequencing to optimize antifungal treatment as early as pos-sible.

DETAILED DESCRIPTION:
The major problem in managing life threatening invasive fungal infections in patients (pts) with acute leukemia and pts after allogeneic hematopoietic stem cell transplantation is the lack of sensitive and specific diagnostic tools to identify fungal pathogens reliably and early in the course of the disease. Because of deep neutropenia and low platelet count, invasive diagnostic procedures are rarely feasible in time, therefore bronchoscopy with BAL is the method of choice in diagnosing pulmonary infections, as the sensitivity of culture-based methods from blood is low, especially in mould infections. Indirect methods, so-called surrogate markers, are becoming increasingly important in this clinical setting. These serologic markers, mainly galactomannan (GM) and recently 1(1,3)-β-D-glucan (BDG), have been validated in clinical trials for blood samples, however the clinical significance of testing BAL samples is up to now only based on retrospective data for GM and has not been reported yet for BDG.

The aim of our prospective and multicentre diagnostic study is therefore to elucidate on the sensitivity and specificity rates of these serologic markers in combination with molecular tools (both an Aspergillus specific and a multifungal PCR based assay), as serologic markers are not pathogen-specific, and furthermore to define species-specific cut-off values for BDG in BAL samples.

Additionally, if genomic material of Aspergillus fumigatus is detected by PCR in a clinical sample, we investigate fungal DNA for point mutations in the cyp51A gene mediating resistance against common mould-active triazoles with novel rapid, sensitive and specific, non-culture-based PCR-assays and sequencing to optimize antifungal treatment as early as possible.

This study aims to improve the early, sensitive and specific diagnosis of invasive pulmonary fungal infections and detect azole resistance patterns, it might impact on the prognosis in hematologic patients; therefore antifungal treatment data and clinical outcome will be recorded.

Clinical samples (BAL and blood) from approximately 100 pts suffering from acute leukemia and pts after allogeneic stem cell transplantation with febrile neutropenia and lung infiltrates diagnosed in a chest CT scan suggestive for fungal infection will be investigated after pts's informed consent in a multicentre, prospective trial. Pts will undergo standardized diagnostic imaging and microbiological procedures for identification of the underlying infectious pathogen. BAL and blood samples will be tested additionally for GM, BDG and with a diagnostic nested Aspergillus PCR assay, a multifungal DNA-Microarray and an azole resistance PCR assay. The molecular assays were established by our group and encompass the detection of Aspergillus fumigatus, Aspergillus flavus, Aspergillus terreus, Candida albicans, Candida dubliniensis, Candida glabrata, Candida lusitaniae, Candida tropicalis, Fusarium oxysporum, Fusarium solani, Mucor racemosus, Rhizopus microsporus, Scedosporium prolificans, Trichosporon asahii and identify the three most common point mutations that confer resistance to triazoles like voriconazole or posaconazole.

Results of other diagnostic means including culture findings as well as patients' clinical data (e.g. duration of neutropenia, underlying disease and outcome including follow-up data concerning antifungal treatment and mortality attributable to fungal infections) will be documented, pseudonomyzed and included in our data bank.

BAL and blood aliquots of 20 control pts without immunosuppression (suffering from lung diseases) will be collected and tested identically.

Case definitions will be made according to 2008 EORTC/MSG criteria. The duration of the study will be approximately 24 months

ELIGIBILITY:
Inclusion Criteria:

* acute leukemia or after allogeneic stem cell transplantation
* febrile neutropenia
* lung infiltrates suggestive for fungal infection (halo sign. nodules, air-crescent sign)

Exclusion Criteria:

* missing informed consent
* other underlying diagnosis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering from acute leukemia and pts after allogeneic stem cell transplantation with febrile neutropenia and lung infiltrates diagnosed in a chest CT scan suggestive for fungal infection will be investigated after pts's informed consent in a multicentre, prospective trial
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-08; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic certainty | 6 Weeks
  After 6 weeks the diagnostic performance of the biomarkers and their combination in relation to diagnostic accuracy will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Buchheidt, MD, Principal Investigator — Medical Faculty Mannheim, University of Heidelberg
Locations (1):
- University Hospital Mannheim, Mannheim, Germany

REFERENCES:
- [Background] Reinwald M, Hummel M, Kovalevskaya E, Spiess B, Heinz WJ, Vehreschild JJ, Schultheis B, Krause SW, Claus B, Suedhoff T, Schwerdtfeger R, Reuter S, Kiehl MG, Hofmann WK, Buchheidt D. Therapy with antifungals decreases the diagnostic performance of PCR for diagnosing invasive aspergillosis in bronchoalveolar lavage samples of patients with haematological malignancies. J Antimicrob Chemother. 2012 Sep;67(9):2260-7. doi: 10.1093/jac/dks208. Epub 2012 Jun 27. PMID 22740590
- [Background] Reinwald M, Spiess B, Heinz WJ, Vehreschild JJ, Lass-Florl C, Kiehl M, Schultheis B, Krause SW, Wolf HH, Bertz H, Maschmeyer G, Hofmann WK, Buchheidt D. Diagnosing pulmonary aspergillosis in patients with hematological malignancies: a multicenter prospective evaluation of an Aspergillus PCR assay and a galactomannan ELISA in bronchoalveolar lavage samples. Eur J Haematol. 2012 Aug;89(2):120-7. doi: 10.1111/j.1600-0609.2012.01806.x. Epub 2012 Jun 22. PMID 22650156
- [Background] Spiess B, Seifarth W, Merker N, Howard SJ, Reinwald M, Dietz A, Hofmann WK, Buchheidt D. Development of novel PCR assays to detect azole resistance-mediating mutations of the Aspergillus fumigatus cyp51A gene in primary clinical samples from neutropenic patients. Antimicrob Agents Chemother. 2012 Jul;56(7):3905-10. doi: 10.1128/AAC.05902-11. Epub 2012 Apr 23. PMID 22526309
- [Derived] Spiess B, Postina P, Reinwald M, Cornely OA, Hamprecht A, Hoenigl M, Lass-Florl C, Rath PM, Steinmann J, Miethke T, Lauten M, Will S, Merker N, Hofmann WK, Buchheidt D. Incidence of Cyp51 A key mutations in Aspergillus fumigatus-a study on primary clinical samples of immunocompromised patients in the period of 1995-2013. PLoS One. 2014 Jul 29;9(7):e103113. doi: 10.1371/journal.pone.0103113. eCollection 2014. PMID 25072733